CLINICAL TRIAL: NCT03355729
Title: The Quebec Family Study: an Observational Study Aimed at Investigating the Role of Genetic Factors in Physical Fitness, Obesity and Risk Factors for Common Diseases and Health-related Behaviours
Brief Title: The Quebec Family Study (QFS): Role of Genetic Factors in Obesity and Its Related Risk Factors and Diseases
Acronym: QFS
Status: Completed | Type: Observational
Sponsor: Louis Pérusse (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Louis Pérusse, Professor, Laval University
Organization: Laval University (Other)
Other Study IDs: 2010-075 CG
Record Dates: First submitted 2017-11-16; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Physical Fitness
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA is available from subjects that were enrolled in Phases 2 and 3 of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Quebec Family Study (QFS) is an observational study that was planned to investigate the role of genetic factors in physical fitness, body composition, risk factors for common disease and health-related behaviour.

DETAILED DESCRIPTION:
The Quebec Family Study was an observational study with three cycles of data collection between 1978 and 1992. During the first cycle of data collection (Phase 1: 1978-1982), a total of 1,650 subjects from 375 families were recruited. During the second cycle (Phase 2: 1989-1997), 385 subjects from 105 phase 1 families were retested and an additional 372 subject from 74 families were recruited. During the third cycle (Phase 3: 1998-2002), 204 subjects from phase 1 were tested a third time, 113 subjects from phase 2 were tested a second time and 194 new subjects from 44 families were recruited.

ELIGIBILITY:
Inclusion Criteria:

* Age over 10 years

Exclusion Criteria:

* Not applicable

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The QFS cohort is a mixture of random sampling and ascertainment through obese individuals. In Phase 1 of the study, subjects were randomly selected from French-Canadian families living in the Quebec city area, In Phases 2 and 3 of the study, families with a least one obese parent and one obese offspring were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 951 (Actual)
Dates: Start 1978-06 (Actual); Primary Completion 2002-09-05 (Actual); Study Completion 2002-09-05 (Actual)

PRIMARY OUTCOMES:
Body composition | Through study completion, an average of 24 years
  Body composition as assessed by underwater weighing
Body mass index (kg/m^2) | Through study completion, an average of 24 years
  Body mass index assessed from height and weight
Abdominal fat | Through study completion, an average of 24 years
  Abdominal fat as assessed by commuted tomography
Waist and hip circumferences (cm) | Through study completion, an average of 24 years
  Waist and hip circumferences (cm)

SECONDARY OUTCOMES:
Caloric intake | Through study completion, an average of 24 years
  Total caloric intake and macronutrient intake using a 3-day dietary record
Eating behaviour | Through study completion, an average of 24 years
  Eating behaviour assessed using the Three-Factor Eating questionnaire
Energy expenditure | Through study completion, an average of 24 years
  Oxygen consumption at rest and during exercise
Physical activity level | Through study completion, an average of 24 years
  Physical activity level assessed by questionnaire
Blood pressure (mm Hg) | Through study completion, an average of 24 years
  Systolic and diastolic blood pressure
Plasma lipid levels (mmol/L) | Through study completion, an average of 24 years
  Fasting levels of triglycerides, LDL-cholesterol and HDL-cholesterol in mmo/L
Glucose levels (mmol/L) | Through study completion, an average of 24 years
  Plasma glucose levels in a fasting state and following an oral glucose tolerance test, inflammatory markers.
  Plasma glucose levels in a fasting state and during an oral glucose tolerance test
Insulin levels (pmol/L) | Through study completion, an average of 24 years
  Plasma insulin levels in a fasting state and following an oral glucose tolerance test.
C-reactive protein (CRP in mg/ml) | Through study completion, an average of 24 years
  C-reactive protein (CRP in mg/ml)
Adiponectin levels (in micrograms/ml) | Through study completion, an average of 24 years
  Adiponectin levels (in micrograms/ml)
Interleukin-6 (IL6) and tumor necrosis factor-alpha (TNF-alpha) in pg/ml | Through study completion, an average of 24 years
  Interleukin-6 (IL6) and tumor necrosis factor-alpha (TNF-alpha) in pg/ml
Smoking habits (nb of cigarettes per day) | Through study completion, an average of 24 years
  Smoking habits (nb of cigarettes per day)
Sleeping (hours/day) | Through study completion, an average of 24 years
  Sleeping (hours/day)
Alcohol consumption | Through study completion, an average of 24 years
  Alcohol consumption (nb of drinks per week)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Bouchard, Ph.D., Principal Investigator — Pennington Biomedical Center; Louis Perusse, Ph.D., Study Director — Laval University

REFERENCES:
- [Background] Chaput JP, Perusse L, Despres JP, Tremblay A, Bouchard C. Findings from the Quebec Family Study on the Etiology of Obesity: Genetics and Environmental Highlights. Curr Obes Rep. 2014 Jan 4;3(1):54-66. doi: 10.1007/s13679-013-0086-3. eCollection 2014. PMID 24533236
- [Derived] Jacob R, Drapeau V, Tremblay A, Provencher V, Bouchard C, Perusse L. The role of eating behavior traits in mediating genetic susceptibility to obesity. Am J Clin Nutr. 2018 Sep 1;108(3):445-452. doi: 10.1093/ajcn/nqy130. PMID 29982344
- See also: PubMed citation — http://www.ncbi.nlm.nih.gov/pubmed/24533236